CLINICAL TRIAL: NCT05835141
Title: Rates and Risk Factors of Contact Between the OTX-TIC Intracameral Ocular Implant and Corneal Endothelium
Status: Completed | Type: Observational
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Benjamin Xu, Assistant Professor, University of Southern California
Other Study IDs: The XU Study
Record Dates: First submitted 2023-04-17; First posted 2023-04-28 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Corneal Endothelium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: OCT Imaging — Each participant will receive imaging of the inferior sectors of the iridocorneal angle at 150°, and 180°, and 210° with the swept-source ANTERION AS-OCT system under standardized light and dark lighting conditions by a trained research technician

SUMMARY:
To determine what proportion of patients have inferior angle recess dimensions that could accommodate the OTX-TIC, and what are risk factors for implant contact with the corneal endothelium.

ELIGIBILITY:
Inclusion Criteria:

* Age over 40 years
* No history of ocular surgery other than cataract surgery

Exclusion Criteria:

- Media opacities that preclude OCT imaging of the anterior segment

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study aims to enroll 100 patients undergoing routine evaluation with Dr. Benjamin Xu at the USC Roski Eye Institute.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-01-30 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
Primary Outcome 1 | 4-6 Months
  Predict contact between simulated OTX-TIC implant and corneal endothelium imaged using the ANTERION AS-OCT system.
Primary Outcome 2 | 4-6 Months
  Characterize the variability in distance (mean and standard deviation) between the angle recess and Schwalbe's line
Primary Outcome 3 | 4-6 Months
  Calculate the proportion of eyes with predicted contact between the simulated implant and corneal endothelium.
Primary Outcome 4 | 4-6 Months
  Develop logistic regression models to identify demographic, clinical, and biometric risk factors for predicted contact.

CONTACTS AND LOCATIONS:
Locations (1):
- USC Roski Eye Institute, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No